CLINICAL TRIAL: NCT06399107
Title: Lentiviral Vector Gene Therapy in Sickle Cell Disease Using Autologous CD34+ Hematopoietic Stem Cells Collected Via Apheresis and Modified With a Lentiviral Vector
Brief Title: Investigation Into the Use of BAH243 Lentiviral Vector for Gene Therapy in Treating Sickle Cell Disease
Acronym: BAH243
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202493
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease; Sickle-Cell Disease With Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Treatment (CD19/BCMA-CAR T cells, chemotherapy) (Experimental): Participants will be administered a one-time dose of the Drug Product, created using their own CD34+ hematopoietic stem cells which are gathered through plerixafor-induced mobilization and apheresis. These cells are then modified with the BAH243 lentiviral vector (LVV), which carries the human beta-A-T87Q globin gene.
  Additionally, the same process of plerixafor mobilization and apheresis will be employed to collect rescue cells.
  Interventions: Genetic: Drug Product is administered by IV infusion following myeloablative conditioning with busulfan

INTERVENTIONS:
Genetic: Drug Product is administered by IV infusion following myeloablative conditioning with busulfan — An autologous CD34+ cell-enriched population from patients with sickle cell disease (SCD), which includes hematopoietic stem cells (HSCs) that have been transduced with the BAH243 lentiviral vector (LVV) carrying the βA-T87Q-globin gene, is preserved in a cryopreservation solution.
  Other Names: BAH243

SUMMARY:
This study is an open-label, non-randomized, single-dose Phase 1/2 trial involving around 85 adult and pediatric participants aged between 2 and 50 years with sickle cell disease (SCD). It aims to assess the effectiveness of hematopoietic stem cell transplantation (HSCT) using BAH243 for SCD.

DETAILED DESCRIPTION:
Participants in this study will be involved for two years following their transplant. Those who join will also be invited to partake in a subsequent long-term follow-up study, which will continue to evaluate the safety and effectiveness of the treatment for an additional 13 years, culminating in a total of 15 years of observation post-infusion of the drug product. This clinical trial is structured as a single-arm, single-dose, single-center, open-label study without any dose escalation involved. Its main goal is to investigate the safety of the study drug in treating sickle cell disease (SCD). The treatment regimen, including myeloablative conditioning, will only commence for subsequent participants once the initial participant has successfully completed dosing and undergone a safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of SCD, with either βS/βS, βS/β0, or βS/β+ genotype.
* Be ≥2 and ≤50 years of age at time of consent.
* Weigh a minimum of 6 kg.
* Have a Karnofsky performance status of ≥60 (≥16 years of age) or a Lansky performance status of ≥60 (<16 years of age).
* Be treated and followed for at least the past 24 months prior to Informed Consent in medical center(s) that maintained detailed records on sickle cell disease history.
* In the setting of appropriate supportive care measures (e.g., pain management plan), have experienced at least 4 protocol-defined VOEs in the 24 months prior to informed consent.
* Have either experienced HU failure at any point in the past or must have intolerance to HU (intolerance is defined as the patient being unable to continue to take HU per PI judgment).
* Female and male subjects of childbearing potential agree to use 1 method of highly effective contraception from Screening to at least 6 months after drug product infusion.
* Provision of written informed consent for this study by subject, or as applicable, subject's parent(s)/legal guardian(s).

Exclusion Criteria:

* Subjects for whom allogeneic hematopoietic stem cell transplantation (allo-HSCT) is medically appropriate per PI judgment and a willing, human leukocyte antigen (HLA)-matched related hematopoietic stem cell donor is available.
* Severe cerebral vasculopathy, defined by any history of overt ischemic or hemorrhagic stroke, a history of abnormal transcranial Doppler (TCD) or TCD imaging (TCDI) for subjects ≤ 16 years of age (e.g. TCD velocity >200 cm/sec) requiring ongoing chronic transfusions, a Screening TCD or TCDI velocity > 200 cm/sec (central read), a Screening MRA showing > 50% stenosis or occlusion in the circle of Willis (central read), or a Screening MRA showing the presence of Moyamoya (central read).
* Positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2), hepatitis B, hepatitis C, human T-lymphotropic virus-1 (HTLV-1), active syphilis.
* Clinically significant, active bacterial, viral, fungal, or parasitic infection
* Advanced liver disease, such as
* clear evidence of liver cirrhosis, active hepatitis or significant fibrosis (based on MRI or liver biopsy)
* liver iron concentration ≥15 mg/g unless liver biopsy shows no evidence of cirrhosis, active hepatitis or significant fibrosis
* Inadequate bone marrow function, as defined by an absolute neutrophil count of <1×10^9/L (<0.5×10^9/L for subjects on hydroxyurea treatment) or a platelet count <100×10^9/L.
* Any contraindications to the use of plerixafor during the mobilization of hematopoietic stem cells and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients.
* Patients needing therapeutic anticoagulation treatment during the period of conditioning through platelet engraftment
* Unable to receive pRBC transfusion.
* Prior receipt of an allogeneic transplant.
* Prior receipt of gene therapy.
* Any prior or current malignancy or immunodeficiency disorder, except previously treated, non-life threatening, cured tumors such as squamous cell carcinoma of the skin.
* Immediate family member with a known or suspected Familial Cancer Syndrome.
* Female subject is breastfeeding, pregnant or will attempt to become pregnant from Screening to at least 6 months after drug product infusion.
* Any other condition that would render the subject ineligible for HSCT.
* Participation in another clinical study with an investigational drug within 30 days of screening.
* Presence of a chromosomal abnormality or genetic mutation that may put the subject at an increased risk of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) per Investigator's judgment.
* Presence of genetic mutations that result in the inactivation of 2 or more α-globin genes

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
VOE-CR | 6-18 months post-transplant
  Proportion of subjects achieving complete resolution of VOEs between 6 months and 18 months after drug product infusion

SECONDARY OUTCOMES:
sVOE-CR | 6-18 months post-transplant
  Proportion of subjects achieving complete resolution of severe vaso-occlusive events, between 6 months and 18 months after drug product infusion
The proportion of subjects achieving Globin Response | 6-24 months post-transplant
  Globin Response, defined as meeting the following criteria for a continuous period of at least 6 months after drug product infusion:
  * Weighted average HbAT87Q percentage of non-transfused total Hb* ≥30% AND
  * Weighted average non-transfused total Hb* increase of ≥3 g/dL compared to baseline total Hb* OR weighted average non-transfused total Hb* ≥10 g/dL
  * non-transfused total Hb is the total g/dL of HbS + HbF + HbA2 + HbAT87Q

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No